CLINICAL TRIAL: NCT00431041
Title: VECTOR: A Randomized Double-blind Study to Assess the Safety and Efficacy of Solifenacin (Vesicare®) in Comparison to Oxybutynin for Overactive Bladder Patients
Brief Title: Study to Compare the Safety and Efficacy of Solifenacin With Oxybutynin for the Treatment of Overactive Bladder (VECTOR)
Acronym: VECTOR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma Canada, Inc. (Industry)
Responsible Party: Sr Manager Clinical Trial Registry, Astellas Pharma US, Inc
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VES-001
Record Dates: First submitted 2007-02-01; First posted 2007-02-02 (Estimated); Results first posted 2010-01-11 (Estimated); Last update posted 2010-06-08 (Estimated); Status verified 2010-06

CONDITIONS: Overactive Bladder
Keywords: Solifenacin succinate; Oxybutynin immediate release; Xerostomia; Overactive bladder
MeSH Terms: conditions — Urinary Bladder, Overactive; Xerostomia | interventions — Solifenacin Succinate; oxybutynin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Solifenacin (Experimental): Solifenacin succinate: 5 mg tablets, taken orally, once daily
  Interventions: Drug: solifenacin
- Oxybutynin IR (Active Comparator): Oxybutynin Immediate Release: 5 mg capsules, taken orally, 3 times a day
  Interventions: Drug: oxybutynin immediate release

INTERVENTIONS:
Drug: solifenacin — Oral
  Other Names: VESIcare®; YM905
  Arms: Solifenacin
Drug: oxybutynin immediate release — Oral
  Arms: Oxybutynin IR

SUMMARY:
The purpose of this study is to compare the safety and efficacy of solifenacin with oxybutynin immediate-release (IR) for the treatment of overactive bladder (OAB).

DETAILED DESCRIPTION:
This study is a prospective randomized, double-blind, double-dummy, multicentre, 2-arm (1 Active, Active Control) comparative parallel group study to compare the safety and efficacy of solifenacin with oxybutynin immediate-release (IR) for the treatment of overactive bladder (OAB).

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years and older.
* Overactive bladder symptoms for greater than or equal to 3 months and as documented in a 3-day patient diary following screening and preceding baseline visit: > 1 urge episodes/24 hours (average); greater than or equal to 8 micturitions/24 hours (average)

Exclusion Criteria:

* Urinary tract infection, chronic inflammation such as interstitial cystitis and bladder stones
* Clinically significant outflow obstruction
* Uncontrolled narrow angle glaucoma, urinary, or gastric retention
* Severe renal or hepatic impairment
* Chronic severe constipation or history of diagnosed GI obstructive disease
* Significant stress incontinence or mixed stress/urge incontinence where stress is the predominant factor
* Diagnosis or history of neurogenic bladder
* History of bladder or pelvic cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2006-12; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Canada, Inc.
Locations (9):
- Canada (9):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - Halifax, Nova Scotia
  - Guelph, Ontario
  - Kitchener, Ontario
  - Toronto, Ontario
  - Montreal, Quebec

REFERENCES:
- [Background] Herschorn S, Stothers L, Carlson K, Egerdie B, Gajewski JB, Pommerville P, Schulz J, Radomski S, Drutz H, Barkin J, Paradiso-Hardy F. Tolerability of 5 mg solifenacin once daily versus 5 mg oxybutynin immediate release 3 times daily: results of the VECTOR trial. J Urol. 2010 May;183(5):1892-8. doi: 10.1016/j.juro.2010.01.012. Epub 2010 Mar 29. PMID 20303119
- [Derived] Herschorn S, Pommerville P, Stothers L, Egerdie B, Gajewski J, Carlson K, Radomski S, Drutz H, Schulz J, Barkin J, Hirshberg E, Corcos J. Tolerability of solifenacin and oxybutynin immediate release in older (> 65 years) and younger (</= 65 years) patients with overactive bladder: sub-analysis from a Canadian, randomized, double-blind study. Curr Med Res Opin. 2011 Feb;27(2):375-82. doi: 10.1185/03007995.2010.541433. Epub 2010 Dec 23. PMID 21175373
- [Derived] Herschorn S, Vicente C, Piwko C. Canadian cost-effectiveness analysis of solifenacin compared to oxybutynin immediate-release in patients with overactive bladder. J Med Econ. 2010;13(3):508-15. doi: 10.3111/13696998.2010.509244. PMID 20690893
- See also: Link to prescribing information — http://www.astellas.com/ca/media/pdf/Vesicare_Product_Monograph.pdf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Solifenacin | Oxybutynin IR
Started | 68 (Data represents Intention To Treat(ITT) Population: All randomized subjects) | 64 (Data represents ITT Population: All randomized subjects)
Completed | 52 | 40
Not Completed | 16 | 24

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Solifenacin | Oxybutynin IR | Total
Number analyzed (Participants) | 68 | 64 | 132
Age, Customized [Number; unit: participants]
  <=65 years | 41 | 34 | 75
  >65 years | 27 | 30 | 57
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 52 | 103
  Male | 17 | 12 | 29
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 62 | 57 | 119
  Black | 2 | 5 | 7
  Asian | 3 | 0 | 3
  Aboriginal | 0 | 1 | 1
  Hispanic | 0 | 0 | 0
  Other | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: The Number of Subjects Reporting Incidence of Dry Mouth as an Adverse Event
Description: The number of subjects reporting incidence of dry mouth as an adverse event (AE) following direct questioning at each patient follow-up visit
Time Frame: 8 weeks
Population: Data represents ITT Population: all randomized subjects
Measure: Number; unit: participants
Arm/Group | Solifenacin | Oxybutynin IR
Number analyzed (Participants) | 68 | 64
participants | 24 | 53
Statistical Analysis 1: Comparison: Solifenacin vs Oxybutynin IR; Test type: Superiority or Other; p < 0.0001, Chi-squared

2. Primary Outcome: The Severity of Dry Mouth Reported as an Adverse Event
Description: The number of subjects reporting dry mouth at each severity level when dry mouth was reported as an Adverse Event (AE).
  Dry mouth severity was categorized as "mild" (relieved with fluid/hard candy), "moderate" (dry mouth and throat with no difficulty swallowing solid food/water) & "severe" (very dry mouth & throat, difficulty swallowing solid food without water)
Time Frame: 8 weeks
Population: Data represents ITT Population: all randomized subjects
Measure: Number; unit: participants
Arm/Group | Solifenacin | Oxybutynin IR
Number analyzed (Participants) | 68 | 64
participants
  Mild | 18 | 16
  Moderate | 3 | 22
  Severe | 3 | 15
Statistical Analysis 1: Comparison: Solifenacin vs Oxybutynin IR; Test type: Superiority or Other; p = 0.0010, Chi-squared — P-value represents overall comparison of severity of dry mouth

3. Secondary Outcome: Change From Baseline in Micturition Frequency as Reported in Subject 3-day Diary
Description: Subjects were instructed to complete the diary in the 3 day period immediately proceding the visit. Subjects recorded each micturition or instance of passing urine in the toliet.
  The mean was calculated for each time point as the average of the day 1-3 measurements from the associated 3 day diary. Change from baseline was calculated as Week 8- Baseline.
Time Frame: Baseline and 8 Weeks
Population: Data represents ITT Population: all randomized subjects. The numbers of subjects for each time point are noted in the category titles. Data for week 8 and Change from Baseline to week 8 includes all subjects who completed the study
Measure: Mean (Standard Deviation); unit: Micturitions per day
Arm/Group | Solifenacin | Oxybutynin IR
Number analyzed (Participants) | 68 | 64
Micturitions per day
  Change in micturition frequency at 8 wks(N=52; 40) | -2.3 (3.3) | -3.1 (2.7)
  Micturition frequency at Baseline (N=68; 64) | 12.4 (3.2) | 12.5 (3.1)
  Micturition frequency at 8 weeks (N=52; 40) | 9.9 (3.7) | 9.0 (2.9)

4. Secondary Outcome: Change From Baseline in Urgency Episodes as Reported in Subject 3-day Diary
Description: Subjects were instructed to complete the diary in the 3 day period immediately preceding the visit. Subjects recorded each urgency episode or instance of strong desire to pass urine.
  The mean was calculated for each time point as the average of the day 1-3 measurements from the associated 3 day diary. Change from Baseline was calculated as Week 8- Baseline.
Time Frame: Baseline and 8 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: urgency episodes per day
Arm/Group | Solifenacin | Oxybutynin IR
Number analyzed (Participants) | 68 | 64
urgency episodes per day
  Change in urgency episodes at 8 weeks (N=52; 40) | -2.65 (4.54) | -3.70 (3.26)
  Urgency episodes at Baseline (N= 68; 64) | 6.3 (3.98) | 6.6 (4.43)
  Urgency episodes at 8 weeks (N=52; 40) | 3.8 (5.04) | 2.1 (2.88)

ADVERSE EVENTS:
Arm/Group | Solifenacin | Oxybutynin IR
Serious Adverse Events (participants affected / at risk) | 3/68 | 0/64
Other Adverse Events (participants affected / at risk) | 36/68 | 56/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Solifenacin (N=68) | Oxybutynin IR (N=64)
fracture, right foot (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cervical adenocarcinoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Worsening depression (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Solifenacin (N=68) | Oxybutynin IR (N=64)
Dry Eye (Eye disorders) | 0 (0) | 3 (3)
Constipation (Gastrointestinal disorders) | 9 (10) | 4 (4)
Dry Mouth (Gastrointestinal disorders) | 24 (25) | 53 (56)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 5 (5)
Fatigue (General disorders) | 4 (4) | 6 (6)
Nasopharyngitis (Infections and infestations) | 0 (0) | 3 (3)
Urinary tract infection (Infections and infestations) | 3 (5) | 3 (3)
Dizziness (Nervous system disorders) | 2 (2) | 6 (6)
Headache (Nervous system disorders) | 2 (2) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (6)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 9 (9)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Somnolence (Nervous system disorders) | 1 (1) | 3 (3)

LIMITATIONS AND CAVEATS:
The relatively high incidence of AEs, specifically dry mouth, in both groups may be a result of the direct questioning methodology used. Subjects were also informed the primary objectives were the relative frequency and severity of dry mouth.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs may not present or publish data prior to publication of the multicenter data or 12 months have elapsed following database lock.

Sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period of up to 90 days from the time submitted to the sponsor for review.

PIs may not engage in contacts with the media related to the study, study interventions or data without prior written consent.